CLINICAL TRIAL: NCT06675448
Title: In Search of Best Practices for Patients With Heart Failure and Secondary Mitral Regurgitation: An Evaluation of the Inova Heart Failure Treatment Algorithm
Status: Recruiting | Type: Observational
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Other Study IDs: U20-09-4258
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Mitral Regurgitation; Valvular Heart Disease; Heart Failure
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Valve Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Moderate MR: Patients who present with moderate MR and remain in this state will be re-evaluated at 6 months by a phone call and EMR review for ConComitant Cardiac Medication Review, NYHA Class and Adverse Event Evaluation. At 12 months a follow-up evaluation that will include a review of medications, NYHA class, KCCQ, 6MWT, BNP, Adverse Event review and TTE.
  Interventions: Other: Moderate MR
- Mitraclip: For patient who undergo Mitraclip, the safety and effectiveness of the procedure will be evaluated and all peri-procedural complications recorded using the same definitions for procedural success and complications used in the COAPT trial
  Interventions: Device: MitraClip

INTERVENTIONS:
Device: MitraClip — Participants will undergo the Mitraclip procedure according to current standards of practice
  Other Names: MitraClip™ System
  Groups: Mitraclip
Other: Moderate MR — Patients who present with moderate MR (Mitral regurgitation) will serve also as an internal control against which the outcomes of Mitraclip treated patients)
  Groups: Moderate MR

SUMMARY:
The overarching goal of this research proposal is to study the feasibility and clinical impact of implementing an Inova system-wide heart failure treatment algorithm for patients with symptomatic heart failure due to reduced left ventricular ejection fraction (HFreF) and secondary MR

Aim is to check the effectiveness of the IHFTA in identifying patients who are most likely to benefit from percutaneous transcatheter Mitraclip repair in real world

DETAILED DESCRIPTION:
All patients passing through the IHFTA will be tracked and followed w.r.t. their final therapies. Monthly meetings will occur with the IHFTA research team to assess and discuss any challenges in implementing the protocol. Impediments will be identified, and strategies put forth to address them. To examine whether the Inova IHFTA identifies the patient most likely to benefit from Mitraclip, the baseline clinical and echocardiographic characteristics of patients treated with Mitraclip within the IHFTA (who would have met the criteria for COAPT study) will be compared to those of the treated cohort in the COAPT trial using t-tests and Chi-squared tests

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic MR (≥2+) due to cardiomyopathy of either ischemic or nonischemic etiology
* Subject has been adequately treated per applicable standards, including for coronary artery disease, LV dysfunction, MR, and HF.
* NYHA functional class II, III, or ambulatory IV
* Local heart team has determined that MV surgery will not be offered as a treatment option even if the subject is randomized to the Control group.
* LVEF ≤50%.
* LVESD ≤70 mm
* The primary regurgitant jet , in the opinion of the MitraClip implanting investigator, can be successfully treated by the MitraClip (if a secondary jet exists, it must be considered clinically insignificant).
* Transseptal catheterization and femoral vein access is feasible per the MitraClip implanting investigator.
* Age 18 y or older
* Subject or guardian agrees to all provisions of the protocol
* NT-proBNP≥ 1500ng/ml or BNP≥ 300ng/ml

Exclusion Criteria:

* Untreated clinically significant coronary artery disease requiring revascularization
* CABG, PCI, or TAVR within the prior 30 d
* Aortic or tricuspid valve disease requiring surgery or transcatheter intervention
* COPD requiring continuous home oxygen therapy or chronic outpatient oral steroid use
* Cerebrovascular accident within prior 30 d
* Severe symptomatic carotid stenosis (N70% by ultrasound)
* Carotid surgery or stenting within prior 30 d
* ACC/AHA stage D HF
* Presence of any of the following:
* Estimated PASP N70 mm Hg assessed by site based on echocardiography or right heart catheterization, unless active vasodilator therapy in the catheterization laboratory is able to reduce the PVR to b3 Wood units or between 3 and 4.5 Wood units with v wave less than twice the mean of the PCWP
* Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing HF other than dilated cardiomyopathy of either ischemic or nonischemic etiology
* Infiltrative cardiomyopathies (eg, amyloidosis, hemochromatosis, sarcoidosis)
* Hemodynamic instability requiring inotropic support or mechanical heart assistance
* Physical evidence of right-sided congestive HF with echocardiographic evidence of moderate or severe right ventricular dysfunction
* Implant of CRT or CRT-D within the last 30 d
* Mitral valve orifice area <4.0 cm2 by site-assessed TTE
* Leaflet anatomy which may preclude MitraClip implantation, proper MitraClip positioning on the leaflets, or sufficient reduction in MR by the MitraClip
* Hemodynamic instability defined as persistent systolic pressure <90 mm Hg with or without afterload reduction, cardiogenic shock, or the need for inotropic support or intra-aortic balloon pump or other hemodynamic support device
* Need for emergent or urgent surgery for any reason or any planned cardiac surgery within the next 12 m
* Life expectancy <12 m due to noncardiac conditions
* Investigators opinion a condition that could limit the subject's participation
* Status 1 heart transplant or prior orthotopic heart transplantation
* Prior mitral valve leaflet surgery or any currently implanted prosthetic mitral valve, or any prior transcatheter mitral valve procedure
* Echocardiographic evidence of intracardiac mass, thrombus, or vegetation
* Active endocarditis or active rheumatic heart disease or leaflets degenerated from rheumatic disease (ie, noncompliant, perforated)
* Active infections requiring current antibiotic therapy
* TEE is contraindicated or high risk
* Known hypersensitivity or contraindication to procedural medications which cannot be adequately managed medically
* Pregnant or planning pregnancy within next 12m
* Currently participating in an investigational drug or another device study that has not reached its primary end point
* Subject belongs to a vulnerable population or has any disorder that compromises his/her ability to give written informed consent and/or to comply with study procedures.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for this study include adult patients > 18 years of age who have symptomatic (NYHA class II-IVa) HFreF due to ischemic or idiopathic dilated cardiomyopathy (LV ejection fraction ≤ 50%), moderate (2+) to severe (4+) secondary MR and either at least 1 HF hospitalization within the prior 12 months or an elevated brain natriuretic peptide (BNP≥300) or N-terminal pro b-type natriuretic peptide (NT-proBNP ≥ 1500) and have been determined by the site's local heart team as not being appropriate for MV surgery. This study population is similar to patients enrolled in COAPT, but includes patients who present with moderate 2+ MR and others who may end up needing only optimal GDMT and/or CRT or Cardiomems.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2029-09-10 (Estimated); Study Completion 2030-09-10 (Estimated)

PRIMARY OUTCOMES:
Change in NYHA from baseline to 6 months in patients who undergo Mitraclip | baseline to 6 months post Mitraclip procedure
  There are 4 levels of NYHA:
  I (Mild): No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, or dyspnea.
  II (Mild): Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea.
  III (Moderate): Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV (Severe): Unable to carry out any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. If any physical activity is undertaken, discomfort is increased. Improvement is defined as moving from a higher numerical NYHA level to a lower numerical NYHA level (e.g., IV to III).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Sherwood, MD, Principal Investigator — Inova Health Care Services
Locations (1):
- Inova Fairfax Medical Campus, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nkomo VT, Gardin JM, Skelton TN, Gottdiener JS, Scott CG, Enriquez-Sarano M. Burden of valvular heart diseases: a population-based study. Lancet. 2006 Sep 16;368(9540):1005-11. doi: 10.1016/S0140-6736(06)69208-8. PMID 16980116
- [Background] Rossi A, Dini FL, Faggiano P, Agricola E, Cicoira M, Frattini S, Simioniuc A, Gullace M, Ghio S, Enriquez-Sarano M, Temporelli PL. Independent prognostic value of functional mitral regurgitation in patients with heart failure. A quantitative analysis of 1256 patients with ischaemic and non-ischaemic dilated cardiomyopathy. Heart. 2011 Oct;97(20):1675-80. doi: 10.1136/hrt.2011.225789. Epub 2011 Jul 31. PMID 21807656
- [Background] Hayashi S, Fushimi H. [Shock and lymphatic circulation]. Nihon Rinsho. 1970 Jan;28(1):84-9. No abstract available. Japanese. PMID 4908819
- [Background] Stone GW, Lindenfeld J, Abraham WT, Kar S, Lim DS, Mishell JM, Whisenant B, Grayburn PA, Rinaldi M, Kapadia SR, Rajagopal V, Sarembock IJ, Brieke A, Marx SO, Cohen DJ, Weissman NJ, Mack MJ; COAPT Investigators. Transcatheter Mitral-Valve Repair in Patients with Heart Failure. N Engl J Med. 2018 Dec 13;379(24):2307-2318. doi: 10.1056/NEJMoa1806640. Epub 2018 Sep 23. PMID 30280640
- [Background] Obadia JF, Messika-Zeitoun D, Leurent G, Iung B, Bonnet G, Piriou N, Lefevre T, Piot C, Rouleau F, Carrie D, Nejjari M, Ohlmann P, Leclercq F, Saint Etienne C, Teiger E, Leroux L, Karam N, Michel N, Gilard M, Donal E, Trochu JN, Cormier B, Armoiry X, Boutitie F, Maucort-Boulch D, Barnel C, Samson G, Guerin P, Vahanian A, Mewton N; MITRA-FR Investigators. Percutaneous Repair or Medical Treatment for Secondary Mitral Regurgitation. N Engl J Med. 2018 Dec 13;379(24):2297-2306. doi: 10.1056/NEJMoa1805374. Epub 2018 Aug 27. PMID 30145927
- [Background] Yurewicz EC, Sacco AG, Subramanian MG. Pathways to immunocontraception: biochemical and immunological properties of glycoprotein antigens of the porcine zona pellucida. Adv Exp Med Biol. 1986;207:407-27. doi: 10.1007/978-1-4613-2255-9_22. PMID 3825685
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):e38-360. doi: 10.1161/CIR.0000000000000350. Epub 2015 Dec 16. No abstract available. PMID 26673558
- [Background] Sahyoun NR, Lentzner H, Hoyert D, Robinson KN. Trends in causes of death among the elderly. Aging Trends. 2001 Mar;(1):1-10. doi: 10.1037/e620692007-001. No abstract available. PMID 11894224
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Oct 15;62(16):e147-239. doi: 10.1016/j.jacc.2013.05.019. Epub 2013 Jun 5. No abstract available. PMID 23747642
- [Background] Larson SL. Trophoblastic disease. Minn Med. 1967 Jan;50(1):81-6. No abstract available. PMID 4292097
- [Background] Golander A, Spirer Z, Bogair N, Konforti N. [Mima polymorpha bacteremia]. Harefuah. 1973 Sep 2;85(5):220-1. No abstract available. Hebrew. PMID 4755414
- [Background] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Background] Mack MJ, Abraham WT, Lindenfeld J, Bolling SF, Feldman TE, Grayburn PA, Kapadia SR, McCarthy PM, Lim DS, Udelson JE, Zile MR, Gammie JS, Gillinov AM, Glower DD, Heimansohn DA, Suri RM, Ellis JT, Shu Y, Kar S, Weissman NJ, Stone GW. Cardiovascular Outcomes Assessment of the MitraClip in Patients with Heart Failure and Secondary Mitral Regurgitation: Design and rationale of the COAPT trial. Am Heart J. 2018 Nov;205:1-11. doi: 10.1016/j.ahj.2018.07.021. Epub 2018 Aug 1. PMID 30134187
- [Background] Green CP, Porter CB, Bresnahan DR, Spertus JA. Development and evaluation of the Kansas City Cardiomyopathy Questionnaire: a new health status measure for heart failure. J Am Coll Cardiol. 2000 Apr;35(5):1245-55. doi: 10.1016/s0735-1097(00)00531-3. PMID 10758967
- [Background] Callaghan P, Brodie J. Laboratory investigation of sewer swabs following the Aberdeen typhoid outbreak of 1964. J Hyg (Lond). 1968 Dec;66(4):489-97. doi: 10.1017/s0022172400028230. No abstract available. PMID 4885562
- [Background] Zotter-Tufaro C, Mascherbauer J, Duca F, Koell B, Aschauer S, Kammerlander AA, Panzenboeck A, Sadushi-Kolici R, Bangert C, Laimer D, Ristl R, Lang IM, Bonderman D. Prognostic Significance and Determinants of the 6-Min Walk Test in Patients With Heart Failure and Preserved Ejection Fraction. JACC Heart Fail. 2015 Jun;3(6):459-466. doi: 10.1016/j.jchf.2015.01.010. PMID 26046839